CLINICAL TRIAL: NCT04041778
Title: Understanding the Electrophysiological Substrate Underlying Persistent Atrial Fibrillation Study II (USURP AF- Study II)'
Brief Title: 'Understanding the Electrophysiological Substrate Underlying Persistent Atrial Fibrillation Study II (USURP AF- Study II)'
Acronym: USURPAF
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0689
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation Mechanisms; Persistent Atrial Fibrillation; Substrate Ablation; Pulmonary Vein Isolation; Non-contact Mapping
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Catheter ablation — Substrate ablation. Pulmonary vein isolation.

SUMMARY:
Atrial fibrillation (AF) is the most common type of chronic heart rhythm disease worldwide, with significant associated co-morbidities. Although there have been advances in understanding the mechanisms of AF, the underlying cause of AF and factors which perpetuate it remain incompletely understood. This is particularly the case for persistent AF (persAF). Drug treatments for persAF have a role but can have undesirable side effects with relatively limited efficacy. Furthermore, current invasive therapies for persAF remain suboptimal, requiring significant resources, and with potentially serious complications for patients.

Catheter ablation is an effective treatment for paroxysmal AF. For persistent AF (persAF), however, catheter ablation does not provide similar results. This is because there remains a poor understanding of the electrophysiological mechanisms driving persAF. Part of this study aims to further explore the specific locations that represent important substrates which would guide more effective catheter ablation. There have been several different ablation approaches explored in the past (see below), however, these did not improve the outcome post procedure compared with pulmonary vein isolation alone. A pilot study has already been carried out and I aim to expand this further with a larger cohort of patients (10-20) over 2 years. In this study the investigators want to explore whether stable high dominant frequency (HDF) sites (with a high organisation index) act as potential drivers of Atrial Fibrillation. Thus, targeting these sites may results in prolongation of the cycle length and thus possible termination of the arrhythmia.

DETAILED DESCRIPTION:
There are an estimated 1.4 million people in the UK with atrial fibrillation (AF), which accounts for 2.4% of the adult population.1 It is well established that AF is a major causative factor for ischaemic stroke and systemic embolism.2 In addition, strokes resulting from AF carry the highest morbidity and mortality of any other form of stroke. AF is also associated with increased morbidity in relation to heart failure.3,4,5 The UK 2016/7 Sentinal Stroke National Audit Programme (SSNAP) reported that in 7,483 patients with known AF who were not anticoagulated before their stroke, there was a 26% mortality and 45% were discharged with moderate-severe disability.6 AF, therefore, is not only associated with increased mortality and morbidity but also significant healthcare costs.

Broadly speaking AF is characterized by a rapid erratic depolarization of the atrial myocardium which manifests clinically as an irregular pulse which can be rapid. This is diagnosed initially on clinical suspicion by palpation of the pulse and then definitively by an ECG which will show irregular intervals between the QRS complex and absence of a P-wave. Clinically patients may be asymptomatic, however typical associated symptoms include palpitations, (exertional) dyspnoea, syncope/presyncope and chest pains. The patient may experience a variation of these symptoms.

The classification of AF is dependent on several factors: presentation, duration and spontaneous termination. There are 5 defined patterns of AF: First diagnosed AF is that which has not been previously diagnosed irrespective of duration and severity of AF-related symptoms. Paroxysmal AF which self terminates, usually within 48 hours. This includes AF episodes which are cardioverted within 7 days. Persistent AF, which lasts longer than 7 days. Long standing persistent AF, continuous AF lasting >1 year when it is decided to adopt a rhythm control strategy. Permanent AF implies that AF has been accepted by both the patient and the physician, therefore there would be no further pursuit of rhythm control intervention. [2016 ESC Guidelines for the management of atrial fibrillation].

The management of AF is two-fold. Where clinically indicated the patient should be anticoagulated. Over the last seven years four non-VKA OACs (NOACs)-dabigatran, a direct thrombin inhibitor and rivaroxaban, apixaban and Edoxaban, factor Xa inhibitors-have been tested against warfarin in large randomised controlled trials.7-10 These NOACs have been shown to be at least as effective as warfarin in stroke prevention, with a superior safety profile, consistently reducing intracranial haemorrhage.11 Other practical advantages of the NOACs include very few drug interactions and a predictable onset and offset that eliminates the requirement for regular anticoagulation monitoring. This has led to the 2014 NICE AF Guideline giving an equal first-line recommendation for NOACs alongside warfarin for stroke prevention.12 NICE also recommends that the options for anticoagulation should be discussed with the patient and the choice should be based on their clinical features and preferences. The second treatment option is pursuit of either a rhythm or rate control strategy. Rate control is achieved via drug therapy. When aiming for rhythm control the option are 1) anti-arrhythmic drugs (AADs) or 2) Invasive catheter ablation.

At present, current AADs have limited efficacy in maintaining sinus rhythm in patients with AF. In addition, there side effect profiles may prevent their long term use in some patients, even where they are maintaining sinus rhythm.13 The most common drug used for maintenance of sinus rhythm is Amiodarone which carries a significant side effect profile. In particular there is a risk posed from long term use of thyroid dysfunction (hyper- or hypothyroidism), liver cirrhosis and lung fibrosis.

Patients who have intolerable symptomatic AF which is not responding to medical therapy can be offered invasive treatment in the form of an ablation. The two methods of ablation are cryoablation and radiofrequency ablation. The procedure is carried out under sedation or general anaesthesia. Catheters are introduced via sheaths placed in the femoral vein and guided up to the right atrium. Catheters are usually placed at the level of the His and CS. The patient is given heparin and a transeptal puncture is performed to gain access to the left atrium. The pulmonary veins are located and radiofrequency energy or the cryoballoon is applied to specific areas of the left atrial myocardium and around the pulmonary veins. The patients cardiac rhythm is monitored via body surface ECGs and intracardiac electrograms (EGMs). Piccini et al published a meta-analysis in 2009 which showed that PVI increased freedom from AF at 1 year, compared with a non-ablation treatment strategy in those patients with paroxysmal AF.14 Outcomes in persAF are less encouraging. Patients may require multiple procedures to gain true symptom control. Catheter ablation is not without it risks. These include Stroke, cardiac tamponade, diaphragmatic paralysis secondary to damage to the phrenic nerve and oesophageal perforation. Appropriate patient selection is therefore incredibly important.

Sustained AF perpetuates further AF. Simply put, this occurs because with sustained AF the atria become fibrosed and therefore exhibit scar. Over time the atria become electrically and structurally remodeled causing further perpetuation of the arrhythmia.

A paper by Haïssaguerre et al. in 1998 showed that when the atria and pulmonary veins were mapped with intracardiac catheters isolated ectopic activity was a trigger for a pAF episode. Theses site then underwent RF ablation. The pulmonary veins were found to be the predominant sites of earliest activation and RF ablation at these sites prevented further pAF.15 Pulmonary vein isolation is now the cornerstone of therapy for patients with symptomatic drug refractory pAF.

A better understanding of the mechanisms of persAF is still needed to improve catheter ablation outcomes. Over the last decade, different ablation approaches have been proposed including i) an anatomical one, with ablation lines mimicking the Cox Maze procedure, and ii) electrical strategies which aim at identifying critical atrial sites with electrical signatures that harbour areas of relevant remodeling believed to perpetuate or drive the chaotic fibrillatory rhythm, whereby their ablation would terminate AF and prevent its induction. Early results appeared promising ablating at sites where the recordings indicated complex fractionated atrial electrograms (CFAEs) and also with a signal processing approach to identify focal and /or rotor activity (FIRM mapping) but these results were proved to be difficult to replicate and a more recent randomised study (STAR-AF II) showed that generic linear and CFAE ablation did not improve the ablation outcome over and above pulmonary vein isolation (PVI) alone.16

Also, heterogeneity in patient characteristics would explain the variable results and precision medicine approaches are needed to design patient specific therapeutic strategies. Better ways to identifying relevant atrial substrate are needed and to demonstrate that targeting these locations improve ablation outcome.

Study Hypothesis

There are specific locations within the atria (left atrium specifically) which exhibit electrical characteristics which act as drivers in persistent atrial fibrillation. These sites can be analysed by non-contact mapping techniques which will more accurately guide catheter ablation.

Proposal

The aim of USURP-II AF is to expand upon the work carried out in USURP-I and that is to be able to determine driver characteristics and mechanisms of persistent atrial fibrillation. The investigators still need to better understand the electrophysiological mechanisms underlying persistent AF so that the investigators can have a guided approach to ablation in persistent AF. Limitations of USURP-I included too shorter data analysis times (30 seconds only from 5 minutes of exported data) purely due to lack of computer processing power. In addition, only centre of gravity of DF clouds were analysed and no comparison of rotor behaviour was done. The latter analysis is now possible. In the original study both prolonging of the cycle length and termination of the arrhythmia were end points in determining successful vs. unsuccessful ablation. Analysis of both DF and rotor behaviour at successful vs. unsuccessful sites in longer recordings would allow refinement of the characteristics and criteria for ablation which the investigators plan to apply prospectively in this new study.

It should be noted that this is not a clinical trial and that I am studying the different mechanisms of PersAF after applying the below ablation strategy, rather than outcomes. The patients recruited will be on a standard care pathway and will not be recruited for the sole purposes of the study. The following is broad overview of the how I intend to carry out the clinical aspect of the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged 18 years or over
* Must be able to communicate in written and spoken English
* Must be able to give signed informed consent.
* All patients must be defined as having persistent atrial fibrillation (AF > 7 days) and must be in AF at the start of the procedure.
* The patient preferably should be undergoing AF ablation for the first time, however repeat ablations can be permitted.
* The patient must be listed for persistent AF ablation as part of standard clinical care.

Exclusion Criteria:

* Symptoms secondary to ischaemic or valvular heart disease
* Congenital heart disease
* Previous history of a cardiac arrhythmia (other than AF, atrial tachycardia, atrial flutter).
* Previous cardiothoracic surgery
* Underlying severe respiratory disease (i.e. patient on long term oxygen therapy)
* Medical conditions which will affect cardiac rhythm, even if treated (e.g. thyroxine, etc.)
* Presence of chest deformity.
* Left atrial dilatation (L or R atrial end-diastolic dimension > 4.5cm in any conventional plane of measurement on 2D transthoracic echocardiography).
* Presence of implantable cardiac defibrillator or pacemaker (including cardiac resynchronisation devices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will have been diagnosed with Persistent Atrial Fibrillation (persAF). They will have been listed for a first time persAF ablation as part of standard routine care.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Termination to sinus rhythm | in procedure
Slowing of cycle length by greater than or equal to 20milliseconds | in procedure
Termination of AF in to an organised atrial tachyarrhythmia | in procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Andre Ng, MBChB, PhD., Principal Investigator — Professor of Electrophysiology University Hospitals Leicester
Locations (1):
- University Hospitals Leicester NHS Foundation Trust, Glenfield Hospital, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No